CLINICAL TRIAL: NCT01273909
Title: Outcomes After Perforator Flap Reconstruction for Breast Reconstruction and/or Lymphedema Treatment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The National Institute of Lymphology (Industry)
Collaborators: The DrMarga Practice Group (Unknown); The Center for Restorative Breast Surgery, LLC (Other)
Responsible Party: Principal Investigator, Marga F. Massey, M.D., Principle Investigator, The National Institute of Lymphology
Other Study IDs: MFM001; 1116697 (Other: Western Institutional Review Board)
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2); Acquired Lymphedema; Congenital Lymphedema
Keywords: Breast Cancer; BRACA1/2 Genotype; Acquired Lymphedema; Congenital Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Perforator Flap Breast Reconstruction: Patients who undergo perforator flap breast reconstruction with or without concomitant vascularized lymph node transfer
  Interventions: Procedure: Perforator Flap Breast Reconstruction; Procedure: Vascularized Lymph Node Transfer
- Vascularized Lymph Node Transfer: Patients who undergo perforator flap vascularized lymph node transfer with or without concomitant perforator flap breast reconstruction
  Interventions: Procedure: Perforator Flap Breast Reconstruction; Procedure: Vascularized Lymph Node Transfer

INTERVENTIONS:
Procedure: Perforator Flap Breast Reconstruction — perforator flap breast reconstruction with or without vascularized lymph node transfer
  Other Names: DIEP Flap; SGAP Flap; IGAP Flap; SIEA Flap; TUG Flap; TDAP Flap; ICP Flap
Procedure: Vascularized Lymph Node Transfer — perforator flap vascularized lymph node transfer with or without concomitant perforator flap breast reconstruction
  Other Names: VLNTx

SUMMARY:
The goal of this prospective, observational study is to investigate the clinical, psychosocial, and patient satisfaction outcomes of patients who undergo perforator flap reconstruction for breast reconstruction and/or vascularized lymph node transfer (VLNTx) for the treatment of lymphedema.

The investigators hypothesize that (1) perforator flap breast reconstruction will result in excellent clinical, psychosocial, and patient satisfaction outcomes compared to non-perforator flap breast reconstruction; (2) perforator flap breast reconstruction is associated with less persistent postsurgical pain than other forms of breast reconstruction, even after controlling for major cofactors, such as the extent of auxiliary lymph node dissection and the use of radiation therapy; (3) perforator flap reconstruction for the treatment of Lymphedema (i.e., VLNTx ) will result in the reduction of symptoms and complications of lymphedema.

DETAILED DESCRIPTION:
Breast cancer is a serious health issue that affects 1 in 8 women. Although numerous treatments have arisen in recent years to aggressively combat this disease and increase survivorship, many survivors develop a crippling condition that can result in devastating physical and psychological impairments. Breast reconstruction by any method may help recovery psychologically. However, some individuals still report experiencing pain following their recovery from surgery. Additionally, secondary lymphedema is a common yet poorly understood complication of breast cancer patients. For those individuals who undergo axillary lymph node dissection the rates of incidence of lymphedema approach 47%. These rates tend to increase further for patients who receive irradiation treatment or mastectomies. Currently there is no known cure for lymphedema. Current treatments include non-invasive measures as well as surgical interventions. Vascularized lymph node transfer (VLNTx) is a fairly recent surgical procedure that has shown promising results.

The goal of this research study is to analyze the clinical outcome of subjects who undergo breast reconstruction with perforator flaps and/or VLNTx using information collected as part of standard care.

Clinical data will be collected prospectively. All subjects who undergo a surgical procedure will complete the online persistent postsurgical pain assessment questionnaire.

The BreastQ questionnaire will be completed by patients prior to and after undergoing breast reconstruction and/or lymphedema treatment.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing perforator flap surgery for breast reconstruction and/or vascularized lymph node transfer for treatment of lymphedema

Exclusion Criteria:

* Pregnant
* unable to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are patients of the "Dr Marga" Practice or the Center for Restorative Breast Surgery that consent to participate in this research study will be selected. There is no age, ethnicity or gender requirement.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in BreastQ Questionnaire and Lymphedema Severity Score | Baseline and 6 months after surgery

SECONDARY OUTCOMES:
Persistent Postsurgical Pain assessment questionnaire | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marga F. Massey, M.D., Principal Investigator — National Institute of Lymphology
Locations (3):
- United States (3):
  - National Institute of Lymphology, Chicago, Illinois
  - The Center for Restorative Breast Surgery, New Orleans, Louisiana
  - The DrMarga Practice Group, Charleston, South Carolina

REFERENCES:
- [Background] Massey MF, Spiegel AJ, Levine JL, Craigie JE, Kline RM, Khoobehi K, Erhard H, Greenspun DT, Allen RJ Jr, Allen RJ Sr; Group for the Advancement of Breast Reconstruction. Perforator flaps: recent experience, current trends, and future directions based on 3974 microsurgical breast reconstructions. Plast Reconstr Surg. 2009 Sep;124(3):737-751. doi: 10.1097/PRS.0b013e3181b17a56. PMID 19730293
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Dayangac M, Makay O, Yeniay L, Aynaci M, Kapkac M, Yilmaz R. Precipitating factors for lymphedema following surgical treatment of breast cancer: implications for patients undergoing axillary lymph node dissection. Breast J. 2009 Mar-Apr;15(2):210-1. doi: 10.1111/j.1524-4741.2009.00703.x. No abstract available. PMID 19292814
- [Background] Becker C, Assouad J, Riquet M, Hidden G. Postmastectomy lymphedema: long-term results following microsurgical lymph node transplantation. Ann Surg. 2006 Mar;243(3):313-5. doi: 10.1097/01.sla.0000201258.10304.16. PMID 16495693
- [Background] Rockson SG, Rivera KK. Estimating the population burden of lymphedema. Ann N Y Acad Sci. 2008;1131:147-54. doi: 10.1196/annals.1413.014. PMID 18519968
- See also: National Institute of Lymphology research web page — http://www.nilymph.com/ongoing-clinical-research.php